CLINICAL TRIAL: NCT01446952
Title: A Phase I Dose-Escalation Study of the Safety and Pharmacokinetics of Vitamin E δ-Tocotrienol Following Single Dose Administration in Healthy Subjects
Brief Title: Vitamin E δ-Tocotrienol (VEDT) Single Dose in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); BioGene Life Science (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MCC-16152
Record Dates: First submitted 2011-09-28; First posted 2011-10-05 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-04

CONDITIONS: Pancreatic Cancer
Keywords: prevention; pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — tocotrienol, delta

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dose Escalation (Experimental): Vitamin E δ-Tocotrienol will be administered orally as a single agent once. Vitamin E δ-Tocotrienol is supplied as 100-mg, 200-mg, and 400-mg capsules.
  Interventions: Drug: Vitamin E δ-Tocotrienol

INTERVENTIONS:
Drug: Vitamin E δ-Tocotrienol — The first cohort will be dosed with δ-tocotrienol at 200 mg. A minimum of 3 participants is planned for each dosing cohort with Vitamin E δ-Tocotrienol dose escalation dependent on safety from prior cohorts.
  Other Names: Delta-tocotrienol

SUMMARY:
This is a Phase 1, open-label, non-randomized, dose-finding, study of Vitamin E δ-Tocotrienol in subjects with resectable pancreatic tumors.

DETAILED DESCRIPTION:
Vitamin E tocotrienols have been shown to exhibit cancer-preventive activities in preclinical studies. Vitamin E tocotrienols are composed of α-, β-, δ-, and γ-tocotrienols. The investigators preclinical studies indicate that δ-tocotrienol possesses the most potent antitumor activity against pancreatic cancer. It is believed that this micronutrient may have a role in the prevention of pancreatic cancer in healthy participants who are at increased risk of developing the disease.

ELIGIBILITY:
Inclusion Criteria:

* The participant is ≥ 18 years old
* The participant has an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.
* The participant has adequate organ function as follows:

  * Serum creatinine ≤ 1.5 mg/dL or calculated creatinine clearance ≥ 60 mL/min.
  * Bilirubin ≤ the institutional upper limits of normal (ULN)
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) to be within institutional normal range.
  * Absolute neutrophil count (ANC) ≥ 1000mm³
  * Platelet count ≥ 100,000/mm³
* The participant has the capability of understanding the informed consent document and has signed the informed consent document.
* Sexually active participants (male and female) must use medically acceptable methods of contraception during the course of the study.
* Female participants of childbearing potential must have a negative pregnancy test at screening.
* Able to understand and comply with the requirements of the protocol.

Exclusion Criteria:

* The participant is receiving investigational therapy (other than the investigational therapy under study).
* The participant has received investigational therapy within 30 days prior to first dose of study drug.
* Patients who are unable to swallow capsules.
* Patients with prior malignancies, other than squamous or basal cell carcinomas, unless disease free for ≥ 5 years.
* The participant has had prior major surgery within 30 days prior to first dose of study drug.
* The participant has active infection or fever >38.5C within 3 days prior to first dose of study drug.
* The participant has uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, hypertension, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* The participant is unable or unwilling to stop taking vitamins, herbal remedies, or nonprescription medications.
* The participant is pregnant or breastfeeding.
* The participant is unable or unwilling to abide by the study protocol or cooperate fully with the investigator or designee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-09; Primary Completion 2012-09 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events | 3 weeks per participant
  The primary objective of this study is to evaluate the safety and tolerability of Vitamin E δ-Tocotrienol and to determine the minimally effective dose (MED) or maximum tolerated dose (MTD) of Vitamin E δ-Tocotrienol administered once. Safety will be assessed by standard clinical findings and laboratory tests. Toxicity grade is defined by the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE)v.4.0. Ninety-five percent confidence intervals may be calculated for selected safety and exploratory variables.

SECONDARY OUTCOMES:
Number of Participants With Pharmacokinetic (PK) Markers of Vitamin E δ-Tocotrienol | 3 weeks per participant
  Pharmacokinetic (PK) markers of Vitamin E δ-Tocotrienol in the plasma, urine, and neoplastic tissue of participants with pancreatic neoplasia. To determine the effects of dose on the plasma pharmacokinetic (PK) of Vitamin E δ-Tocotrienol when orally administered as a single dose in healthy subjects. Ninety-five percent confidence intervals may be calculated for selected safety and exploratory variables. Dose escalation will be based on safety and available PK data.
Number of Participants With Pharmacodynamic (PD) Markers of Vitamin E δ-Tocotrienol | 3 weeks per participant
  Pharmacodynamic (PD) Markers of Vitamin E δ-Tocotrienol in the plasma, urine, and neoplastic tissue of participants with pancreatic neoplasia. To evaluate pharmacodynamic (PD) markers of Vitamin E δ-Tocotrienol activity in peripheral blood. Ninety-five percent confidence intervals may be calculated for selected safety and exploratory variables. Correlative analysis of PD data will be done.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Klapman, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States